CLINICAL TRIAL: NCT05646823
Title: A Probiotic Blend in the Improvement of Gastrointestinal Symptoms and Life Quality in Patients With Celiac Disease
Brief Title: Probiotic Blend for Celiac Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Collaborators: Alexandre Faraco (Unknown)
Responsible Party: Principal Investigator, Monique Michels, PhD, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UESCatarinense
Record Dates: First submitted 2022-11-17; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Celiac Disease
Keywords: probiotic; gastrointestinal symptoms; life quality
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): vehicle only - Maltodextrin gluten free
  Interventions: Dietary Supplement: Placebo
- Treatment (Experimental): Bifidobacterium longum CCT 1934; Bifidobacterium lactis CCT 7858; Lactobacillus rhamnosus CCT 7863; Streptococcus thermophilus ATCC 19258) Final concentration: 1 x 10e10 CFU/ day
  Interventions: Dietary Supplement: Probiotic blend

INTERVENTIONS:
Dietary Supplement: Probiotic blend — Bifidobacterium longum CCT 1934; Bifidobacterium lactis CCT 7858; Lactobacillus rhamnosus CCT 7863; Streptococcus thermophilus ATCC 19258) Final concentration: 1 x 10e10 CFU/ day
  Arms: Treatment
Dietary Supplement: Placebo — vehicle only - Maltodextrin gluten free
  Arms: Placebo

SUMMARY:
The objective of the study is to develop a probiotic product (B. longum CCT 1934; B. lactis CCT 7858; L. rhamnosus CCT 7863; S. thermophilus ATCC 19258) to reduce the symptoms caused by celiac disease and concomitantly improve the quality of life of patients. To achieve the objective, 118 volunteers of both sexes will be included, randomly distributed into two groups: Test group (n=59): Volunteers supplemented with the probiotic product (Bifidobacterium longum CCT 1934; Bifidobacterium lactis CCT 7858; Lactobacillus rhamnosus CCT 7863 ; Streptococcus thermophilus ATCC 19258) Final concentration: 1 x 1010 CFU/ day) and Placebo group (n=59): Volunteers supplemented with placebo. The study will be conducted with patients diagnosed with celiac disease, the audience is adults (18 - 65 years old). The study will last for 90 days and volunteers will be invited to participate in three visits. During these visits, participants will be invited to answer the proposed questionnaires. The volunteer is expected to show improvement in gastrointestinal symptoms, as well as an improvement in quality of life after using the probiotic blend for 90 days.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled study to evaluate the effectiveness of a probiotic blend (Bifidobacterium longum CCT 1934; Bifidobacterium lactis CCT 7858; Lactobacillus rhamnosus CCT 7863; Streptococcus thermophilus ATCC 19258) in improving gastrointestinal symptoms caused by celiac disease, as well as improvement in quality of life. Study will be conducted with patients diagnosed with celiac disease by the gastroenterologist participating in the study. Adult audience (18 - 65 years old). In the present study, 118 volunteers of both sexes will be included, randomly distributed into two groups. They will be randomized into: 1) Probiotics: (Bifidobacterium longum CCT 1934; Bifidobacterium lactis CCT 7858; Lactobacillus rhamnosus CCT 7863; Streptococcus thermophilus ATCC 19258) Final concentration: 1 x 1010 CFU/day. 2)Placebo: Capsules containing the gluten-free product vehicle. The study will last for 90 daysVisit 1 (day 0) - Assessment of inclusion and exclusion criteria, clinical and physical evaluation, research presentation and signing of the Free Consent Form and Clarified in writing, partial delivery of the test product or placebo, delivery and application of questionnaires (quality of life questionnaires (CD-QOL scale) and Gastrointestinal Symptom Rating Scale (GSRS) questionnaire for gastrointestinal evaluation. The questionnaires will preferably be applied in a in person by the researchers involved (with scheduled time) in interview format, or online via Google Forms (if the volunteer so prefers), to be agreed with the volunteer. will follow the guidelines according to CIRCULAR LETTER No. 2/2021/CONEP/SECNS/MS, providing confidentiality to all information collected.

In addition, an explanation will also be given on the first visit regarding the importance of the questionnaires, correct completion, and possible changes in the GIT in the first days of using the probiotic. Visit 2 (day 45) - Clinical consultation with a specialist physician, delivery final product test or placebo, and application of questionnaires.Visit 3 (day 90) - Clinical consultation with specialist physician and application of final questionnaires. Closure of the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Free and Informed Consent in writing, signed and dated;
* Age according to the indicated population;
* Patients diagnosed with celiac disease by a specialist physician.

Exclusion Criteria:

* History of daily consumption of probiotics, fermented milk and or yogurt;
* subjects known to have demonstrated a prior reaction, including anaphylaxis, to any substance in the composition of the study product;
* Subjects who have uncompensated blood pressure;
* history of heart disease, including valvular heart disease or any implantable device;
* subjects with active, uncontrolled bowel disease such as Crohn's disease or ulcerative colitis;
* another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-04-17 (Estimated)

PRIMARY OUTCOMES:
gastrointestinal symptom | 12 weeks
  The GSRS is a disease-specific instrument. The 15 items combine into five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The reliability and validity of the GSRS are well-documented, and norm values for a general population are available

SECONDARY OUTCOMES:
Life quality | 12 weeks
  coeliac disease (CD)-related quality of life (QOL) test. CD-QOL has 20 items across four clinically relevant subscales (Limitations, Dysphoria, Health Concerns, and Inadequate Treatment). The CD-QOL has high internal consistency, reliability, and psychometric validation indicates both convergent and discriminate validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Extremo Sul Catarinense, Criciúma, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No
Only this study